CLINICAL TRIAL: NCT00848588
Title: A Survey of Factors Associated With the Successful Recognition of Agonal Breathing and Cardiac Arrest by 9-1-1 Call Takers.
Brief Title: A Survey of Factors Associated With the Successful Recognition of Agonal Breathing and Cardiac Arrest.
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Other Study IDs: PLP 6566
Record Dates: First submitted 2009-02-19; First posted 2009-02-20 (Estimated); Results first posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2022-11

CONDITIONS: Cardiac Arrest
Keywords: agonal breathing; cardiac arrest; 9-1-1 call taker; survey
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Full and part-time 9-1-1 call takers employed at Ambulance Communication Centres in the Canadian provinces of Ontario, Nova Scotia, New Brunswick, as well as the city of Montreal, Quebec, Canada.

SUMMARY:
The overall goal of this pilot study is to design and conduct a survey of 9-1-1 call takers in the province of Ontario, Canada to better understand the factors associated with the successful identification of cardiac arrest (including victims with agonal breathing) over the phone. Specific objectives are:

1. To conduct iterative semi-structured interviews to identify behavioural factors influencing identification of cardiac arrest by 9-1-1 call takers;
2. To develop a survey instrument about behavioural factors influencing the ability of 9-1-1 call takers to identify cardiac arrest based on a systematic review of the literature, the results of the semi-structured interviews, and theoretical constructs from the Theory of Planned Behaviour; and
3. To conduct a survey among Ontario 9-1-1 call takers using the survey instrument, and to identify factors and strategies that might be targeted by Knowledge Translation interventions.

ELIGIBILITY:
Inclusion Criteria:

* 9-1-1 call-takers, male or female, full or part-time, employed in an eligible Ambulance Communication Centre

Exclusion Criteria:

* Ambulance Communication Centre Managers, support staff or administrative staff

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The survey will be sent to all full-time and part-time 9-1-1 call takers employed in the Canadian provinces of Ontario, Nova Scotia and New Brunswick, as well as the city of Montreal, Quebec, Canada.
Sampling Method: Probability Sample
Enrollment: 404 (Actual)
Dates: Start 2009-06; Primary Completion 2010-04 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christian Vaillancourt, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (1):
- Ottawa Hospital Research Institute, Ottawa, Ontario, Canada

REFERENCES:
- [Derived] Vaillancourt C, Jensen JL, Grimshaw J, Brehaut JC, Charette M, Kasaboski A, Osmond M, Wells GA, Stiell IG. A survey of factors associated with the successful recognition of agonal breathing and cardiac arrest by 9-1-1 call takers: design and methodology. BMC Emerg Med. 2009 Jul 31;9:14. doi: 10.1186/1471-227X-9-14. PMID 19646269

RESULTS

PARTICIPANT FLOW:
Groups:
- Survey Respondents: Full and part-time 9-1-1 call takers employed at Ambulance Communication Centres in the Canadian provinces of Ontario, Nova Scotia, New Brunswick, as well as the city of Montreal, Quebec, Canada.
Period: Overall Study
Arm/Group | Survey Respondents
Started | 404
Completed | 404
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Survey Respondents
Number analyzed (Participants) | 404
Age, Continuous [Mean (Full Range); unit: years] | 36.9 [22 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 262
  Male | 142
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Canada | 404

OUTCOME MEASURES:

1. Primary Outcome: Intention to Give CPR Instructions
Description: Median intention to give CPR instructions when agonal breathing is present
Time Frame: During a call with a victim potentially in cardiac arrest
Population: Median intention to give CPR instructions to a caller reporting a victim in cardiac arrest when agonal breathing is present (scale 0-5; 5 is highest)
Measure: Median (Standard Deviation); unit: score on a scale
Arm/Group | Survey Respondents
Number analyzed (Participants) | 404
score on a scale | 4.3 (1.17)

ADVERSE EVENTS:
Arm/Group | Survey Respondents
All-Cause Mortality (participants affected / at risk) | 0/404
Serious Adverse Events (participants affected / at risk) | 0/404
Other Adverse Events (participants affected / at risk) | 0/404

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No